CLINICAL TRIAL: NCT06331494
Title: Efficacy of Butylphthalide on Symptomatic Atherosclerotic Stenosis in Middle Cerebral Artery (SICAS): a Prospective, Randomized, Double-blinded, Placebo-controlled, Multiple-center Trial.
Brief Title: Efficacy of Butylphthalide on Symptomatic Atherosclerotic Stenosis in Middle Cerebral Artery
Acronym: SICAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SICAS
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke, Acute; Intracranial Atherosclerosis
Keywords: dl-3-n-Butylphthalide; atherosclerotic stenosis; middle cerebral artery; stroke
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide (Experimental): The Butylphthalide group will receive Butylphthalide Sodium Chloride injection (100ml, twice/day) for the initial 10±3 days, followed by oral Butylphthalide soft capsules (0.2g, triple/day) for day 11±3 to day 180.
  Interventions: Drug: Butylphthalide
- Placebo (Placebo Comparator): The Placebo group will receive Butylphthalide Placebo injection (100ml, twice/day) for the initial 10±3 days, followed by oral Butylphthalide Placebo soft capsules (0.2g, triple/day) for day 11±3 to day 180.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Butylphthalide — Butylphthalide Sodium Chloride injection for 10±3 days, oral Butylphthalide soft capsules for day 11±3 to day 180.
  Other Names: DL-3-n-butylphthalide
  Arms: Butylphthalide
Drug: Placebo — Butylphthalide Placebo injection for 10±3 days, oral Butylphthalide Placebo soft capsules for day 11±3 to day 180.
  Other Names: Blank
  Arms: Placebo

SUMMARY:
Ischemic stroke with high incidence, mortality, disability and recurrence rate, has become the leading threat to the health worldwide. Intracranial atherosclerotic stenosis (ICAS) is commonly associated with ischemic stroke, especially in Chinese residents. Patients with severe ICAS are subject to a very high risk of recurrent stroke events, despite best medical therapy available. Unstable or complex atherosclerotic plaques can lead to plaque ruptures and distal embolisms, thereby increasing the risk of ischemic stroke recurrence. Studies have shown that activation of inflammatory states may play a driving role in the formation and development of atherosclerosis. So far, it remains unclear which are the best treatments for this condition, especially for high-risk patients. Dl-3-n-butylphthalide (NBP) is a Class I novel drug independently developed in China and was officially approved for use in acute ischemic stroke. Preclinical data showed that NBP can act multiple effects of anti-inflammation, antioxidation and anti-apoptosis by suppressing pro-inflammatory factors and upregulating the expression of anti-inflammatory factors. It is still undetermined whether combined therapy with NBP could enhance the curative effect of intracranial atherosclerosis. The primary purpose of this trial is to evaluate the efficacy of butylphthalide in reducing the degree of arterial stenosis and stabilizing plaques in patients with severe symptomatic middle cerebral artery stenosis.

DETAILED DESCRIPTION:
The SICAS trial is a prospective, randomized, double-blinded, placebo- controlled, multiple-center trial to evaluate the efficacy of butylphthalide in the reduction of symptomatic atherosclerotic stenosis of middle cerebral artery in acute ischemic stroke patients. A total of approximately 140 patients within 7 days of symptom onset of acute ischemic stroke or transient ischemic attack (TIA) will be enrolled. The participants fulfilling the inclusion criteria will be randomized 1:1 into two groups: 1) the Butylphthalide group will receive Butylphthalide Sodium Chloride injection (100ml, twice/day) for the initial 10±3 days, followed by oral Butylphthalide soft capsules (0.2g, triple/day) from day 11±3 to day 180. 2) the Placebo group will receive Butylphthalide Placebo injection (100ml, twice/day) for the initial 10±3 days, followed by oral Butylphthalide Placebo soft capsules (0.2g, triple/day) from day 11±3 to day 180. The study consists of four visits including the day of randomization, day 10±3 when the injection therapy is done, and 90 and 180 days when the oral therapy is finished. The primary end point is the change in degree of atherosclerotic stenosis in the symptomatic middle cerebral artery at 180 days. The atherosclerotic stenosis is evaluated by high-resolution MRI vessel-wall imaging technique. The second end point are rate of recurrence of ischemic stroke or TIA in the qualifying artery within 180 days, the changes in plaque volumes, hemorrhage and enhancement volumes of atherosclerotic plaque in the symptomatic middle cerebral artery, National Institutes of Health Stroke Scale (NIHSS), modified Rankin Scale (mRS), change in cerebral perfusion and concentrations of serum lipid profiles within 180 days.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 55-75 years;
2. At least one of the following risk factors of atherosclerosis: hypertension, diabetes, hypercholesterolemia, or smoking;
3. Symptomatic atherosclerotic stenosis in middle cerebral artery: large artery atherosclerotic cerebral infarction or TIA within 7 days of onset; 70%-99% stenosis of the responsible middle cerebral artery [M1] confirmed by high-resolution MRI examination (referred to Warfarin-Aspirin Symptomatic Intracranial Disease standard); new-onset infarction confirmed by diffusion weighted imaging (DWI) or TIA symptoms in the territory of the responsible artery supply;
4. NIHSS ≤ 20;
5. mRS ≤ 2 at randomization (pre-morbid historical assessment);
6. Participants understand the purpose of the study and have signed informed consent form.

Exclusion Criteria:

1. Presence of intracranial hemorrhage or other pathological brain diseases;
2. Plan to or have performed intravenous thrombolysis or mechanical thrombectomy therapy;
3. Unable to undergo MRI examination;
4. Use Butylphthalide during onset between randomization;
5. Suspect of cardiac embolism, such as atrial fibrillation, artificial heart valves, endocarditis, etc;
6. Contraindications for the use of clopidogrel or aspirin;
7. Known allergy history of celery or butylphthalide;
8. Severe liver dysfunction (aspartate aminotransferase or alanine transaminase > 2 times normal upper limit) or severe renal dysfunction (creatinine value > 1.5 times normal upper limit), heart failure, asthma, etc;
9. History of intracranial hemorrhage, coagulation disorders, systemic bleeding, thrombocytopenia, or other hematological disorders;
10. Plan to perform other surgical procedures or interventional treatments that may require termination of investigational drug use;
11. Severe non-cerebrovascular diseases with an expected survival time less than 3 months;
12. Actively participating in another drug or device trial;
13. Use any drugs with the same or similar mechanism as Butylphthalide during the follow-up period;
14. Unsuitable for this trial from the opinion of the investigators.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in stenosis degree in the responsible artery | 180 days
  Intracranial atherosclerosis is evaluated by high-resolution MRI vessel-wall imaging technique.

SECONDARY OUTCOMES:
Stroke recurrence | 180 days
  Rate of new-onset ischemic stroke or TIA in the territory of the symptomatic middle cerebral artery within 180 days.
Change in plaque volumes the responsible artery | 90 days, 180 days
  Change in plaque volumes in the symptomatic middle cerebral artery at 90 days and 180 days.
Changes in hemorrhage and enhancement volumes of atherosclerotic plaque in the responsible artery | 90 days, 180 days
  Changes in hemorrhage and enhancement volumes of atherosclerotic plaque in the symptomatic middle cerebral artery at 90 days and 180 days.
Changes in National Institutes of Health Stroke Scale (NIHSS) | 10±3 days
  National Institutes of Health Stroke Scale (NIHSS, range: 0 - 42) at baseline and discharge.
Proportion of patients with modified Rankin Scale score (mRS) 0-2 | 90 days, 180 days
  Proportion of patients with modified Rankin Scale score (mRS) 0-2 at 90 days and 180 days.
Change in the value of cerebral blood flow (CBF) in the responsible artery territory | 90 days, 180 days
  Qualitative analysis of regional cerebral blood flow (CBF) in arterial spin labeling sequence in the territory of the symptomatic middle cerebral artery at baseline, 90 days and 180 days.
Change in concentrations of serum lipid profiles | 10±3 days, 90 days, 180 days
  Concentrations of total cholesterol, serum triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol at baseline, discharge, 90 days and 180 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zeng, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No